CLINICAL TRIAL: NCT05962359
Title: Neural Prediction to Enhance Language Outcomes in Children With Cochlear Implant
Brief Title: Neural Prediction to Enhance Language
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Chinese University of Hong Kong (Other); Northwestern University (Other); University of North Carolina, Chapel Hill (Other); University of Southern California (Other); University of Miami (Other); The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Nancy Young, MD, Head, Section of Otology/Neurotology and Medical Director, Audiology & Cochlear Implant Programs, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DC019387 (NIH)
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Bilateral Sensorineural Hearing Loss; Speech and Language Development Delay Due to Hearing Loss; Social Communication
Keywords: Hearing Loss; Children; Parent-mediated intervention; Language prediction
MeSH Terms: conditions — Speech; Communication; Hearing Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-treatment Model Building (No Intervention)
- Communication Treatment (Experimental)
  Interventions: Behavioral: Parent-Implemented Communication Treatment

INTERVENTIONS:
Behavioral: Parent-Implemented Communication Treatment — The intervention will be taught by a qualified professional online and/or in-person for about 6 months. Parents will learn strategies to enhance their children's social communication and will receive coaching and feedback.
  Arms: Communication Treatment

SUMMARY:
The language outcome of children receiving cochlear implantation to address bilateral sensorineural hearing loss is more variable than that of typical hearing children. The research is focused upon development of neural predictive models based upon brain imaging to forecast language after cochlear implantation on the individual child level. The long-term goal is improving children's language by using predictive models to enable a custom "predict to prescribe" approach to intervene with more effective behavioral therapy for children at risk to develop poorer language. The investigators previously developed models for short term language outcome of English-learning implanted children. The aims of this study are to 1. Develop models able to predict long term outcome for English- learning and Spanish-learning children; and 2. To evaluate whether English-learning children predicted to achieve lower language based on the investigators' previously constructed models can demonstrate significant gains from Parent Implemented Communication Treatment (PICT). PICT is an intensive parent education program about strategies to improve children's communication.

DETAILED DESCRIPTION:
Arm1: Non-treatment Model Building. Up to 700 children will be recruited from 5 cochlear implant programs in the United States. Children will be enrolled and followed for up to four years after implantation. Study information will be obtained from each child's medical record before and after implantation including cause of hearing loss, general health, language and communication history, family history, cochlear implant device and surgery. Audiological information before and after implantation will be collected from routine visits that are part of cochlear implant candidacy evaluation and audiology evaluations after implantation. This includes audiology evaluations after activation of the cochlear implant that take place at around 6, 12, 18, 24, 36 and/or 48 months. Pre-surgical MRI done at each participating site as part of routine pre-operative evaluation will also be collected for analysis. If enrolled into the study at Lurie Children's Hospital of Chicago before the pre-surgical MRI is done, the parent or guardian will have the option to have their child undergo additional research scans during the pre-surgical MRI.

Parents will be asked to complete baseline and follow-up surveys. The surveys will ask about family demographic and health information, language exposure in the home, therapy and school services, and language and communication ability of the child. Parental surveys will be readministered at about 12-month intervals after the child's device is turned on. In addition, surveys about the child's cognition will be sent to parents after their child has used their implant for one and two years. Surveys will be offered online by a secure link provided during clinical visits, emailed after the visit or sent by MyChart to the parent/guardian for completion at home.

An in-person research-only speech and language evaluation will be done at about one-year intervals after initial implantation during each year the child is enrolled in the study. The evaluation will take less than two hours.

Arm 2: Communication Treatment. In addition to all of the study procedures described above for Arm1, at only Lurie Children's Hospital of Chicago, 10 children will be enrolled in each of four years who meet additional inclusion criteria. Children enrolled in this arm will receive Parent Implemented Communication Treatment (PICT). PICT involves training parents to use communication skills to support development of their child's language. PICT will consist of one-hour weekly sessions for about six months provided virtually by a secure video chat system such as Zoom. The child and parent/caregiver will both participate in each weekly session. In addition, parent and child social interactions will be evaluated by video chat each month for six months and then annually for two years. The parent and child social interaction evaluation will take less than 15 minutes. Children who receive PICT will continue to receive all other therapies. In other words, no therapies will be discontinued during the time children are receiving PICT.

ELIGIBILITY:
Inclusion Criteria (Arm 1):

1. Children with sensorineural hearing loss who meet clinical criteria for cochlear implantation in both ears who meet the following age criteria at time cochlear implant evaluation begins:

   * Age 5 years and under.
   * English or Spanish as the dominant language.
2. English or Spanish dominant language in the home.

Inclusion Criteria (Arm 2):

1. Children with bilateral sensorineural hearing loss who meet clinical criterial for cochlear implantation
2. English dominant spoken language by family
3. Age at implantation of 36 months and younger when treatment begins
4. Parent or caregiver that is willing to participate who understands spoken English
5. Child is exposed to spoken language by at least one parent (total communication or auditory/oral) in the home

Exclusion Criteria (Arm 1):

1. Severe motor and /or cognitive disability that would preclude evaluation of progress
2. Limited electrode insertion likely to significantly impact development of speech perception
3. Hearing loss due to bacterial meningitis
4. Neither English or Spanish as the dominant family language in the home

Exclusion Criteria (Arm 2):

1. Severe motor and /or cognitive disability that would preclude evaluation of progress
2. Limited electrode insertion likely to significantly impact development of speech perception
3. Hearing loss due to bacterial meningitis
4. Dominant language other than English
5. Diagnoses or medical conditions expected to impact language development independent of hearing loss
6. Cochlear nerve deficiency in implanted ears or severe cochlear malformation
7. Children already having spoken language who score better than 25th percentile on the Words and Sentences portion of the CDI language evaluation.
8. Child with more than two months CI experience prior to start of treatment

Ages: 0 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2027-07-23 (Estimated); Study Completion 2028-01-23 (Estimated)

PRIMARY OUTCOMES:
Preschool Language Scales, Fifth Edition (PLS-5) | At 12 months after cochlear implant activation
  A standardized measure of auditory comprehension and expressive communication in children. Standard scores are obtained which are then translated to percentiles, and age equivalents. Higher standard scores indicate better performance.
Preschool Language Scales, Fifth Edition (PLS-5) | At 24 months after cochlear implant activation
  A standardized measure of auditory comprehension and expressive communication in children. Standard scores are obtained which are then translated to percentiles, and age equivalents. Higher standard scores indicate better performance.
Preschool Language Scales, Fifth Edition (PLS-5) | At 36 months after cochlear implant activation
  A standardized measure of auditory comprehension and expressive communication in children. Standard scores are obtained which are then translated to percentiles, and age equivalents. Higher standard scores indicate better performance.
Preschool Language Scales, Fifth Edition (PLS-5) | At 48 months after cochlear implant activation
  A standardized measure of auditory comprehension and expressive communication in children. Standard scores are obtained which are then translated to percentiles, and age equivalents. Higher standard scores indicate better performance.
Expressive One-Word Picture Vocabulary Test, Fourth Edition (EOWPVT-4) | At 12 months after cochlear implant activation
  An individually administered, norm-referenced assessment of how well a person can name objects, actions, or concepts presented in full-color pictures. Raw scores are obtained which are then translated to standard scores, percentiles, and age equivalents. Both higher standard scores and raw scores indicate better performance.
Expressive One-Word Picture Vocabulary Test, Fourth Edition (EOWPVT-4) | At 24 months after cochlear implant activation
  An individually administered, norm-referenced assessment of how well a person can name objects, actions, or concepts presented in full-color pictures. Raw scores are obtained which are then translated to standard scores, percentiles, and age equivalents. Both higher standard scores and raw scores indicate better performance.
Expressive One-Word Picture Vocabulary Test, Fourth Edition (EOWPVT-4) | At 36 months after cochlear implant activation
  An individually administered, norm-referenced assessment of how well a person can name objects, actions, or concepts presented in full-color pictures. Raw scores are obtained which are then translated to standard scores, percentiles, and age equivalents. Both higher standard scores and raw scores indicate better performance.
Expressive One-Word Picture Vocabulary Test, Fourth Edition (EOWPVT-4) | At 48 months after cochlear implant activation
  An individually administered, norm-referenced assessment of how well a person can name objects, actions, or concepts presented in full-color pictures. Raw scores are obtained which are then translated to standard scores, percentiles, and age equivalents. Both higher standard scores and raw scores indicate better performance.
MacArthur-Bates Communicative Development Inventory (CDI) | At 12 months after cochlear implant activation
  A set of online parent report intruments that evaluate children's early speech and langauge development. Standard scores are based on percentiles for age and sex and range from 1 to 99th percentile. Higher standard scores indicate better performance.
MacArthur-Bates Communicative Development Inventory (CDI) | At 24 months after cochlear implant activation
  A set of online parent report intruments that evaluate children's early speech and langauge development. Standard scores are based on percentiles for age and sex and range from 1 to 99th percentile. Higher standard scores indicate better performance.
MacArthur-Bates Communicative Development Inventory (CDI) | At 36 months after cochlear implant activation
  A set of online parent report intruments that evaluate children's early speech and langauge development. Standard scores are based on percentiles for age and sex and range from 1 to 99th percentile. Higher standard scores indicate better performance.
MacArthur-Bates Communicative Development Inventory (CDI) | At 48 months after cochlear implant activation
  A set of online parent report intruments that evaluate children's early speech and langauge development. Standard scores are based on percentiles for age and sex and range from 1 to 99th percentile. Higher standard scores indicate better performance.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF) | At 12 months after cochlear implant activation
  A parent-reported executive function questionnaire that utilizes T-scores to reflect individual's level of executive functioning. Higher T-scores indicate better performance.
Behavior Rating Inventory of Executive Function (BRIEF) | At 24 months after cochlear implant activation
  A parent-reported executive function questionnaire that utilizes T-scores to reflect individual's level of executive functioning. Higher T-scores indicate better performance.
Behavior Rating Inventory of Executive Function - Preschool Version (BRIEF-P) | At 12 months after cochlear implant activation
  A parent-reported executive function questionnaire designed for preschool-aged children that utilizes T-scores to reflect children's level of executive functioning. Higher T-scores indicate better performance.
Behavior Rating Inventory of Executive Function - Preschool Version (BRIEF-P) | At 24 months after cochlear implant activation
  A parent-reported executive function questionnaire designed for preschool-aged children that utilizes T-scores to reflect children's level of executive functioning. Higher T-scores indicate better performance.
Pediatric Minimum Speech Test Battery (PMSTB) | At 6 months after cochlear implant activation
  A set of measures designed to evaluate speech discrimination for infants and word/ sentence recognition for children using hearing technology before entering school. Scores range from 0 to 700. Higher scores indicate better performance.
Pediatric Minimum Speech Test Battery (PMSTB) | At 12 months after cochlear implant activation
  A set of measures designed to evaluate speech discrimination for infants and word/ sentence recognition for children using hearing technology before entering school. Scores range from 0 to 700. Higher scores indicate better performance.
Pediatric Minimum Speech Test Battery (PMSTB) | At 18 months after cochlear implant activation
  A set of measures designed to evaluate speech discrimination for infants and word/ sentence recognition for children using hearing technology before entering school. Scores range from 0 to 700. Higher scores indicate better performance.
Pediatric Minimum Speech Test Battery (PMSTB) | At 24 months after cochlear implant activation
  A set of measures designed to evaluate speech discrimination for infants and word/ sentence recognition for children using hearing technology before entering school. Scores range from 0 to 700. Higher scores indicate better performance.
Pediatric Minimum Speech Test Battery (PMSTB) | At 36 months after cochlear implant activation
  A set of measures designed to evaluate speech discrimination for infants and word/ sentence recognition for children using hearing technology before entering school. Scores range from 0 to 700. Higher scores indicate better performance.
Pediatric Minimum Speech Test Battery (PMSTB) | At 48 months after cochlear implant activation
  A set of measures designed to evaluate speech discrimination for infants and word/ sentence recognition for children using hearing technology before entering school. Scores range from 0 to 700. Higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Young, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form: Arm 1 - Non-treatment Model Building (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05962359/ICF_000.pdf
  • Informed Consent Form: Arm 2 - Communication Treatment (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05962359/ICF_001.pdf